CLINICAL TRIAL: NCT00529178
Title: A Multicenter, Randomized, Double-blind, Placebo Controlled, Parallel Study to Determine the Efficacy and Safety of Pravastatin 80 mg Administered Once Daily to Hypercholesterolemic Subjects With Chronic, Well Compensated Liver Disease
Brief Title: Pravastatin Efficacy and Safety Trial in Hypercholesterolemic Patients With Chronic Liver Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV123-246
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pravastatin

SUMMARY:
To determine in hypercholesterolemic subjects with chronic, well-compensated liver disease, the percent change from baseline to Week 12 in serum LDL-C of pravastatin 80 mg compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Chronic, well-compensated stable liver
* Hypercholesterolemia

Exclusion Criteria:

* Signs or symptoms of ascites, jaundice, or cirrhosis with a Child-Pugh Score > 5
* History of disorders affecting serum bilirubin levels, more than 1 chronic liver disease, significant endocrine, renal, or gastrointestinal disease, or uncontrolled hypertension
* Treatment with lipid-lowering drugs, unless they have been withdrawn within the timeframe specified in the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2002-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
serum LDL-C | at week 12
ALT value

SECONDARY OUTCOMES:
change in HDL-C, TC and TG | at week 12
clinical symptoms related to acute hepatic injury

REFERENCES:
- [Derived] Lewis JH, Mortensen ME, Zweig S, Fusco MJ, Medoff JR, Belder R; Pravastatin in Chronic Liver Disease Study Investigators. Efficacy and safety of high-dose pravastatin in hypercholesterolemic patients with well-compensated chronic liver disease: Results of a prospective, randomized, double-blind, placebo-controlled, multicenter trial. Hepatology. 2007 Nov;46(5):1453-63. doi: 10.1002/hep.21848. PMID 17668878